CLINICAL TRIAL: NCT01673516
Title: Effect of Renal Sympathetic Denervation on Resistant Hypertension and Cardiovascular Hemodynamic in Comparison to Intensive Medical Therapy Utilizing Impedance Cardiography
Acronym: OsloRDN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/145/REK
Record Dates: First submitted 2012-08-17; First posted 2012-08-28 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Renal sympathetic denervation; Impedance cardiography
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group Co (Active Comparator): group Co receives intensive medical therapy utilizing integrated hemodynamic management calculated by impedance cardiography of "The HOTMAN® System"
  Interventions: Device: The HOTMAN® System
- group RDN (Active Comparator): For patients who will be randomly assigned to undergo renal denervation by "The SymplicityTM Renal Denervation System", the femoral artery will be accessed with the standard endovascular technique and the catheter will be advanced into the renal artery and connected to a radiofrequency generator. As in Symplicity HTN 1 and 2 trials, four-to-six discrete, low-power radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to four-six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm.
  Interventions: Procedure: The SymplicityTM Renal Denervation System

INTERVENTIONS:
Procedure: The SymplicityTM Renal Denervation System — For patients who will be randomly assigned to undergo renal denervation (group RDN), the femoral artery will be accessed with the standard endovascular technique and the catheter will be advanced into the renal artery and connected to a radiofrequency generator. As in Simplicity HTN 1 and 2 trials, four-to-six discrete, low-power radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to four-six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm.
  Arms: group RDN
Device: The HOTMAN® System — Impedance Cardiography by HOTMAN system will evaluates non-invasively hemodynamic parameters in patients randomized to "group Co"
  Arms: group Co

SUMMARY:
The purpose of this study is to demonstrate that Renal Sympathetic Denervation (RDN) improves the control of blood pressure (BP) in patients with treatment-resistant hypertension, as compared to intensive medical therapy (IMT) using hemodynamic parameters and then applying a predefined algorithm of drug selection (i.e. integrated hemodynamic management - IHM) during 6 months intensive treatment program (receiving antihypertensive care according to the 2007 ESH Guidelines). Working hypothesis: When it is possible to disrupt the sympatho-renal axis by RDN - BP reduction occurs to a greater extent and more rapidly than applying intensive medical therapy using IHM.

DETAILED DESCRIPTION:
Hypertension is the most common cardiovascular disease, affecting approximately 1 billion1 people worldwide. Hypertension is a major public health concern, because of its complications (coronary artery disease, heart failure, renal disease, stroke). Early blood pressure control in hypertensive patients guarantees the best prevention of cardiovascular events on the long term (2007 ESH-ESC Guidelines on the Management of Hypertension; VALUE study). However, in spite of education efforts and antihypertensive drugs, blood pressure control rates remain low. The most common cause of uncontrolled BP is inadequate pharmacological treatment, because the selection of antihypertensive agents is often done independently of the hemodynamic status of the patient (volemic status, peripheral resistance, cardiac inotropy).

The sympatho-renal axis describes the dual role of the kidney as originator of some central nervous system afferent signals and recipient of efferent sympathetic signals. Both the contribution of the kidney to central sympathetic drive and the consequences of sympathetic efferent drive to the kidney contribute to the development and sustenance of hypertension. Poly-pharmacy strategies for the treatment of elevated blood pressure have identified populations of patients with treatment resistant hypertension.

Treatment Resistant Hypertension(TRH) is a blood pressure that remains above goal in spite of the concomitant use of antihypertensive medications from more than 3 drug classes. Patients who require more than 4 drug classes to have their blood pressure controlled are also considered to have resistant hypertension. Preferably, the regimen should include a diuretic and all doses should be optimal2 .The true prevalence of treatment resistant hypertension is unknown. In clinical trials from 20 to 40% of randomized patients did not reach blood pressure targets3. In the National Health and Nutrition Examination Survey in USA (2003-2008), non-pregnant adults with hypertension were classified as resistant if their blood pressure was 140/90 mmHg or higher and if they reported using antihypertensive medications from 3 different drug classes or drugs from 4 antihypertensive drug classes regardless of blood pressure. The prevalence was 12.8% of the drug-treated hypertensive population. Risk factors for treatment-resistant hypertension include older age and obesity .

Treatment-resistant patients are more likely to have albuminuria, reduced renal function, and a history of diabetes mellitus, coronary heart disease, stroke or heart failure. They are at increased risk of cardiovascular complications although the true incidence of death and morbidity remains currently unknown.

In the Spanish Ambulatory Blood Pressure Monitoring Registry5, 8295 of 68045 treated patients (12.2%) had treatment resistant hypertension, defined as an office blood pressure equal to or exceeding 140 mm Hg systolic and/or 90 mm Hg diastolic.

RDN is a novel procedure which has been approved safe and gives a remarkable reduction of BP in treatment-resistant hypertensive patients. The HOTMAN® System is a novel impedance cardiographic device, measuring and calculating hemodynamic parameters. The HOTMAN® System may help the physician to control blood pressure in patients with resistance hypertension.

* Our pilot study(Renal sympathetic denervation in patients with treatment-resistant hypertension after witnessed intake of medication before qualifying ambulatory blood pressure.Fadl Elmula FE, Hoffmann P, Fossum E, Brekke M, Gjønnæss E, Hjørnholm U, Kjær VN, Rostrup M, Kjeldsen SE, Os I, Stenehjem AE, Høieggen A.Hypertension. 2013 Sep;62(3):526-32)has showed that The mean office and ambulatory BPs remained unchanged at 1, 3, and 6 months in the 6 patients, whereas there was no known change in antihypertensive medication. Two patients, however, had a fall in both office and ambulatory BPs. Our findings question whether BP falls in response to RDN in patients with true treatment-resistant hypertension.That is why we intended to do an intrim analysis after inclusion of around 30% of the total number planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Average SBP >140mmHg, measured per guidelines
* 24 hour average ABPM daytime SBP >135mm/Hg
* On stable medication regimen of full tolerated doses of 3 or more antihypertensive meds, with one being a diuretic
* No changes for a minimum of 2 weeks prior to screening
* No planned medication changes for 6 months
* Age 18-80 years
* At minimum, 3 antihypertensive medications must meet one or more of the following full dose criteria:
* Highest labeled dose according to medication's labeling
* Highest usual dose per clinical guidelines-JNC-7
* Highest tolerated dose
* Highest appropriate dose for the patient per the PI's clinical judgment

Exclusion Criteria:

* Hemodynamically or anatomically significant renal artery abnormalities or stenosis >50% or prior renal artery intervention
* eGFR < 45 mL/min/1.73m2 (MDRD formula)
* Albumin/creatinine ratio > 50 mg/mmol
* Type 1 diabetes mellitus
* Known alcohol or drug abuse
* Symptomatic orthostatic hypotension in past year
* Stenotic valvular heart disease for which BP reduction would be hazardous
* MI, unstable angina, or CVA in the prior 6 months
* Known primary pulmonary HTN
* Known pheochromocytoma, Cushing's disease, coarctation of the aorta, hyperthyroidism or hyperparathyroidism
* Known primary hyperaldosteronism not adequately treated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Absolute change in office systolic blood pressure(SBP) | at 6 months
  is the absolute change in office SBP, after a 6 months follow-up.

SECONDARY OUTCOMES:
Short and long term safety of RDN as an interventional procedure | up to10 years
  Safety of RDN will be assessed at 1, 3, 5 and 10 years by clinical, laboratory and radiology examinations.
Percentage of normalization of blood pressure(BP) at office, home and ABPM | at 6 months and later
  This will include the percentage of normalization of daytime SBP at office, home and ABPM.
The normalization of hemodynamics. | at 6 month and later
  The normalization of hemodynamics: Cardiac Index (CI), Heart rate, Stroke systemic vascular resistance index (SSVRI), pulse wave velocity(PWV) and central BP.
Cost effectiveness | At 6 month and later
  It will be assessed the Cost effectiveness of Renal denervation as treatment of resistant hypertension compared to control group.

OTHER OUTCOMES:
The quality of life and side effects related to antihypertensive agents | at 6 months and later
  The quality of life and side effects related to antihypertensive agents

CONTACTS AND LOCATIONS:
Overall Officials: Aud Høieggen, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Halvorsen LV, Bergland OU, Soraas CL, Larstorp ACK, Hjornholm U, Kjaer VN, Kringen MK, Clasen PE, Haldsrud R, Kjeldsen SE, Rostrup M, Fadl Elmula FEM, Opdal MS, Hoieggen A. Nonadherence by Serum Drug Analyses in Resistant Hypertension: 7-Year Follow-Up of Patients Considered Adherent by Directly Observed Therapy. J Am Heart Assoc. 2022 Sep 20;11(18):e025879. doi: 10.1161/JAHA.121.025879. Epub 2022 Sep 8. PMID 36073648
- [Derived] Undrum Bergland O, Larstorp ACK, Lund Soraas C, Hoieggen A, Rostrup M, Norheim Kjaer V, Godang K, Sevre K, Fadl Elmula FEM. Changes in sympathetic nervous system activity after renal denervation: results from the randomised Oslo RDN study. Blood Press. 2021 Jun;30(3):154-164. doi: 10.1080/08037051.2020.1868286. Epub 2021 Jan 5. PMID 33399016
- [Derived] Fadl Elmula FE, Hoffmann P, Larstorp AC, Fossum E, Brekke M, Kjeldsen SE, Gjonnaess E, Hjornholm U, Kjaer VN, Rostrup M, Os I, Stenehjem A, Hoieggen A. Adjusted drug treatment is superior to renal sympathetic denervation in patients with true treatment-resistant hypertension. Hypertension. 2014 May;63(5):991-9. doi: 10.1161/HYPERTENSIONAHA.114.03246. Epub 2014 Mar 3. PMID 24591332
- [Derived] Kjeldsen SE, Narkiewicz K, Oparil S, Hedner T. Blood pressure lowering effect of renal sympathetic denervation or placebo? - building expectations for Symplicity-HTN 3. Blood Press. 2013 Oct;22(5):279-81. doi: 10.3109/08037051.2013.840445. No abstract available. PMID 24059787
- [Derived] Fadl Elmula FE, Hoffmann P, Fossum E, Brekke M, Gjonnaess E, Hjornholm U, Kjaer VN, Rostrup M, Kjeldsen SE, Os I, Stenehjem AE, Hoieggen A. Renal sympathetic denervation in patients with treatment-resistant hypertension after witnessed intake of medication before qualifying ambulatory blood pressure. Hypertension. 2013 Sep;62(3):526-32. doi: 10.1161/HYPERTENSIONAHA.113.01452. Epub 2013 Jul 8. PMID 23836798